CLINICAL TRIAL: NCT01409629
Title: Influence of a Computer Game on Youth's Choices of Activities
Status: Terminated | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Sarah-Jeanne Salvy, Assistant Proffessor, University at Buffalo
Other Study IDs: 4325
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Study Individuals' Activity Choices After Playing a Computer Game

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Activity choices: Observe individuals' activity choices after playing a computer game.
  Interventions: Behavioral: Computer game

INTERVENTIONS:
Behavioral: Computer game — Participants will play a computer game

SUMMARY:
Study of activity choices after playing a computer game.

ELIGIBILITY:
Inclusion Criteria:

* Like study foods, healthy

Exclusion Criteria:

* Medical conditions, psychological disorders, food allergies

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy adolescents ages 12-14
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Behavioral Medicine, Buffalo, New York, United States